CLINICAL TRIAL: NCT03971578
Title: Screening Device for Autism Spectrum Disorders Using High Stimulation Rate ABR With Continuous Loop Averaging Deconvolution
Brief Title: Screening for Autism Spectrum Disorders Using Auditory Brainstem Responses
Status: Completed | Type: Observational
Sponsor: Intelligent Hearing Systems (Industry)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Other Study IDs: ASDCLAD001
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Autism Spectrum Disorders Group: Children identified as having Autism Spectrum Disorder Age: 3.5 to 4.5 years old
  Interventions: Other: No Intervention Provided
- Normal Control Group: Normal children without Autism Spectrum Disorder or other identified developmental disability Age: 3.5 to 4.5 years old
  Interventions: Other: No Intervention Provided

INTERVENTIONS:
Other: No Intervention Provided — No Intervention Provided

SUMMARY:
The purpose of this study is to develop an Auditory Brainstem Response (ABR) based neurological screening method to detect increased risk for Autism Spectrum Disorders (ASD) and other neurological conditions in newborns.

DETAILED DESCRIPTION:
In the proposed study, a screening method for neurological deficits, with an emphasis on its application to ASD, will be developed and its feasibility demonstrated. The proposed method will utilize high rate stimulation to acquire Auditory Brainstem Responses in order to determine peak latency and amplitude differences in children with ASD compared to non-ASD. Similarly to newborn hearing screening, the output of the screening method will provide an automated pass or refer outcome that can be used by a physician to determine if the child needs further evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Children with autism spectrum disorder diagnosis
* Normally developing age- and gender-matched controls

Exclusion Criteria:

* Permanent or temporary hearing loss at the time of testing.
* Craniofacial abnormalities

Ages: 42 Months to 54 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with autism spectrum disorders and normally developing age- and gender-matched controls
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami Department of Psychology, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Summary data will be disseminated

REFERENCES:
- [Background] Miron O, Beam AL, Kohane IS. Auditory brainstem response in infants and children with autism spectrum disorder: A meta-analysis of wave V. Autism Res. 2018 Feb;11(2):355-363. doi: 10.1002/aur.1886. Epub 2017 Oct 31. PMID 29087045

RESULTS

PARTICIPANT FLOW:
Groups:
- Autism Spectrum Disorders Group: Children identified as having Autism Spectrum Disorder Age: 2.5 to 7 years old
  No Intervention Provided: No Intervention Provided
- Normal Control Group: Normal children without Autism Spectrum Disorder or other identified developmental disability Age: 2.5 to 7 years old
  No Intervention Provided: No Intervention Provided
Period: Overall Study
Arm/Group | Autism Spectrum Disorders Group | Normal Control Group
Started | 25 | 56
Completed | 14 | 37
Not Completed | 11 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Autism Spectrum Disorders Group | Normal Control Group | Total
Number analyzed (Participants) | 25 | 56 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25 | 56 | 81
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 53.0 (14.2) | 47.3 (17.1) | 49.1 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 28 | 34
  Male | 19 | 28 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 20 | 40 | 60
  More than one race | 2 | 7 | 9
  Unknown or Not Reported | 1 | 5 | 6
Region of Enrollment [Number; unit: participants]
  United States | 25 | 56 | 81

OUTCOME MEASURES:

1. Primary Outcome: ABR Peak V Latency
Description: Auditory Brainstem Response (ABR) peak V latency measurement for the five stimulation rates used in the study. The latency is the time, measured in ms, from the onset of the stimulus to the generation of the response peak component. ABR peak V is the most prominent response peak component in humans.
Time Frame: One Week
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Autism Spectrum Disorders Group | Normal Control Group
Number analyzed (Participants) | 14 | 37
ms
  Peak V Latency at 19.3 Hz Rate | 6 (0.27) | 5.8 (0.16)
  Peak V Latency at 39.3 Hz Rate | 6.29 (0.36) | 5.99 (0.16)
  Peak V Latency at 58.59 Hz Rate | 6.48 (0.25) | 6.26 (0.21)
  Peak V Latency at 195.31 Hz Rate | 7.07 (0.31) | 6.89 (0.25)
  Peak V Latency at 234.38 Hz Rate | 7.45 (0.58) | 7.28 (0.32)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Autism Spectrum Disorders Group | Normal Control Group
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/37
Other Adverse Events (participants affected / at risk) | 0/14 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT03971578/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-30): https://cdn.clinicaltrials.gov/large-docs/78/NCT03971578/SAP_001.pdf
  • Informed Consent Form (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT03971578/ICF_002.pdf